CLINICAL TRIAL: NCT03010111
Title: Latent Tuberculosis Infection in Korean Health Care Workers Using Interferon Gamma Releasing Assay
Brief Title: Latent Tuberculosis Infection in Korean Health Care Workers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hanyang University (Other)
Responsible Party: Principal Investigator, Dong Won Park, assistant professor, Hanyang University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: HYUMC_CM_001
Record Dates: First submitted 2016-12-17; First posted 2017-01-04 (Estimated); Last update posted 2017-01-04 (Estimated); Status verified 2017-01

CONDITIONS: Latent Tuberculosis
Keywords: Latent Tuberculosis; Interferons; Tuberculosis; Healthcare
MeSH Terms: conditions — Latent Tuberculosis; Tuberculosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- health care workers (Other): health care workers including doctors, nurses, technicians and orderly who were hired in 2016 at the Hanyang University Hospital
  Interventions: Other: QFT-IT Test and other blood sampling

INTERVENTIONS:
Other: QFT-IT Test and other blood sampling — In all enrolled health care workers, QFT-IT Test and other blood sampling were performed.

SUMMARY:
The investigators aim to study the prevalence of latent tuberculosis infection (LTBI) using whole-blood interferon-r release assays, and determine the risk factors of LTBI in Korean health care workers.

DETAILED DESCRIPTION:
Further study details as provided by Hanyang University Hospital

ELIGIBILITY:
Inclusion Criteria:

* Health care workers in University affiliated hospital
* Adult aged 20-65

Exclusion Criteria:

* Active tuberculosis
* Subjects diagnosed with HIV infection, malignancy
* Subjects having immunosuppressive drug therapy

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2016-12; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of latent tuberculosis infection developed in Korean health care workers | Three months
  The participants performed QuaniFERON-TB Gold In-Tube test (QFT-IT test) and blood sampling at enrollment. So, the length of time which from the start of the first test of very first participants to the end of test of very last participant is 3 months. The percentage of participants with LTBI in health care workers was evaluated.

SECONDARY OUTCOMES:
Annual incidence of latent tuberculosis infection in Korean health care workers | 1 year after first QFT-IT test (12-15 months)
  QFT-IT test was performed at enrollment and repeated at point of one year after enrollment. So, the length of time which from the start of the first test of very first participants to the end of the second test of very last participant is 12 to 15 months. The percentage of participants with positive conversion in follow-up QFT-IT test (second test) was evaluated in participants who had negative results in the first QFT-IT test. Annual infection of LTBI was evaluated with the conversion of QFT-IT test through annual check up of QFT-IT test.

CONTACTS AND LOCATIONS:
Overall Officials: Jang Won Shon, M.D., Ph.D., Principal Investigator — Hanyang University Hospital, Seoul, Korea
Locations (1):
- Hanyang University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No